CLINICAL TRIAL: NCT03812016
Title: Comparison of Treatment Outcomes for Blepharoptosis of Various Etiologies Using a Feedback-enabled Magnetic Device
Brief Title: A Feedback-enabled Magnetic Device for Temporary Management of Blepharoptosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Collaborators: National Yang Ming Chiao Tung University (Other); The Industrial Technology Research Institute (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Lien, Ching-Feng, Deputy head of the Department of Otolaryngology-Head and Neck Surgery, E-Da Hospital, E-DA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDAHP107026
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Blepharoptosis; Device Usability
Keywords: Blepharoptosis; Blink restoration; Magnetic device; Oculomotor nerve palsy; Ptosis
MeSH Terms: conditions — Blepharoptosis; Oculomotor Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determine device feasibility (Experimental): by evaluating efficacy and safety of the device. Test the device (duration: 120 mins/each time). Intervention: using the feedback-enabled magnetic device.
  Interventions: Device: Feedback-enabled magnetic device

INTERVENTIONS:
Device: Feedback-enabled magnetic device — The device comprises 1 or 2 matched pairs of one near-infrared light-emitting diode and one sensor, a magnetic actuator, an iron sheet, and a biosignal acquisition module. The efficacy and safety were assessed using the feedback-enabled magnetic device.

SUMMARY:
To develop a feedback-enabled magnetic device for management of blepharoptosis and evaluate its efficacy and safety, including the gain of palpebral fissure height, visual field obstruction, blurred vision, foreign body sensation over the cornea, burning or hot sensation over facial skin, and erythema or pruritus over the eyelid, by performing a human trial on patients with blepharoptosis.

DETAILED DESCRIPTION:
The feedback-enabled magnetic device primarily comprises 2 matched pairs of one near-infrared light-emitting diode and one photodiode sensor, a magnetic actuator, an iron sheet (for affixing to the paralytic upper eyelid), and a biosignal acquisition module along with a power supply unit providing a wired connection with optical sensors and a magnetic actuator. Before the study, the differences between the affected and unaffected palpebral fissure heights were directly measured using a ruler. During the test after using the device, the distance of the paralytic eyelid lift was documented and the corrected distance (gain) of the paralytic upper eyelid was calculated. The efficacy and safety of the device were assessed. The efficacy was evaluated according to the symmetrical blinks and gain of paralytic eyelid lifts. Subjective sensation and complications were assessed by visual field obstruction, blurred vision, foreign body sensation over the cornea, burning or hot sensation over facial skin, and erythema or pruritus over the eyelid. After the completion of the study procedure, the eyelid skin integrity, subjective sensation and discomfort were examined. Outcomes in the management of blepharoptosis of diverse etiologies using a feedback-enabled magnetic device will be demonstrated. Differences in outcomes between patients managed using the device and those who underwent surgery will be presented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ptosis; they are capable of understanding and complying with protocol requirements
* Aged 18 years old or older

Exclusion Criteria:

* Upper eyelid scar, contracture, or fibrosis due to previous surgical intervention(s)
* Patients with psychiatric (or mental) disorders; they are unable to cooperate or follow the study procedure
* Children younger than 18 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy by measuring changes in distance. | 10-minutes after completion of the device testing.
  The investigators assess changes (in millimeter) of palpebral fissure height and visual field obstruction before any intervention and during the device intervention by a ruler and a software.
Evaluate visual field changes and discomfort of blurred vision, cornea, upper eyelid, and skin before and after the device use based on a 3-point Likert scale. | 10-minutes after completion of the device testing
  The investigators score questionnaires by assessing visual field changes and discomfort of blurred vision, foreign body sensation over the cornea, burning or hot sensation over facial skin, and erythema or pruritus over the eyelid after device use. According to concepts from the 3-point Likert scale, the scale ranges from 1 to 3 with score 3 indicating no discomfort, score 2 mild to moderate discomfort, and score 1 severe discomfort.
Evaluate frontalis muscle use by measuring changes in muscle activities in both amplitude and fluctuation. | 10-minutes after completion of the testing
  The investigators assess electrical activities of the frontalis muscle and calculate total electromyographic areas (sum of all areas under the curve) before and after the device intervention.

SECONDARY OUTCOMES:
Evaluate the efficacy by measuring changes in distance 1 month and 6 months after surgical intervention. | 1 month and 6 months after completion of surgical intervention.
  The investigators assess changes (in millimeter) of palpebral fissure height and visual field obstruction after surgical intervention (performed after completion of the device intervention) by a ruler and a software.
Evaluate visual field changes and complications 1 month and 6 months after surgical intervention based on a 3-point Likert scale. | 1 month and 6 months after surgical intervention
  The investigators score questionnaires by assessing visual field changes and complications (including cosmetic results, headache relief, undercorrection, infection, foreign body tissue reaction, lagophthalmos, and keratitis). For visual field changes based on the 3-point Likert scale, the scale ranges from 1 to 3 with score 3 indicating good outcomes, score 2 fair outcomes, and score 1 poor outcomes; for complications, with score 3 indicating no discomfort (satisfied), score 2 mild to moderate discomfort (somewhat satisfied), and score 1 severe discomfort (dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Kun Tu, Study Chair — E-Da Hospital, Kaohsiung, Taiwan
Locations (2):
- Taiwan (2):
  - E-Da Hospital, Kaohsiung City
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lien CF, Lin BS, Wu TM, Lin YC, Chang RC, Cheng CK, Yeh JH, Jeng SF. Efficacy and Safety of a Magnetic Device for Temporary Management of Blepharoptosis: Single-Arm Open-Label Trial. Otolaryngol Head Neck Surg. 2025 Nov;173(5):1111-1120. doi: 10.1002/ohn.1350. Epub 2025 Jul 16. PMID 40671431